CLINICAL TRIAL: NCT05640843
Title: A Randomized Placebo Controlled Study of a Plant-Based Dietary Versus Supplement Versus Placebo Intervention in Patients With Monoclonal Gammopathy of Undetermined Significance (MGUS) and Smoldering Multiple Myeloma (SMM) - The Nutrition Prevention (NUTRIVENTION-3) Study
Brief Title: A Study Comparing a Plant-Based Diet With Supplements and Placebo in People With Monoclonal Gammopathy of Undetermined Significance (MGUS) or Smoldering Multiple Myeloma (SMM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Paula and Rodger Riney Foundation (Unknown); Plantable (Unknown); M and M labs (Unknown); VeggieDoctor (Unknown); Sabinsa pharmaceuticals (Unknown); Daily Harvest (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-175
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
Keywords: Plant-Based Diet; Supplements; 22-175
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: This is a randomized, multi-center pilot study with 150 patients (50 per arm). Randomization will be stratified based on BMI and MGUS/SMM status. Randomization in the supplement and placebo arms will be blinded.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily Harvest weekly (Experimental): For 12 weeks, on the Daily Harvest weekly arm, patients will receive two premade meals per day, for lunch and dinner for 6 days weekly, prepared and shipped by U.S.-based company Daily Harvest weekly.
  Interventions: Other: Whole Foods Plant-based Diet
- Supplements (Experimental): For 12 weeks on the supplement arm, patients will be given algae omega 3 supplements (QWell pharmaceuticals) and curcumin supplements (Sabinsa pharmaceuticals) twice daily.
  Interventions: Dietary Supplement: Algae Omega 3 + Curcumin
- Placebo (Placebo Comparator): For 12 weeks on the placebo arm, patients will be given placebo supplements twice daily (QWell and Sabinsa pharmaceuticals).
  Interventions: Other: Placebo supplements

INTERVENTIONS:
Other: Whole Foods Plant-based Diet — The meals will have a low glycemic index and contain legumes, vegetables, whole grains, and plant-based fats that have undergone minimal processing. Detailed recommendations for snacks and breakfasts meeting the standard of a WFPBD will also be given to supplement their daily calorie needs with access to education materials. Patients will also receive dietary education and counselling from a research dietitian every 4 weeks for the 12-week intervention period. They will have access to the team for questions and support as needed
  Arms: Daily Harvest weekly
Dietary Supplement: Algae Omega 3 + Curcumin — For 52 weeks on the supplement arm, patients will be given algae omega 3 supplements and curcumin supplements (Sabinsa pharmaceuticals) twice daily
  Arms: Supplements
Other: Placebo supplements — For 25 weeks on the placebo arm, patients will be given placebo supplements twice daily (Veggie Doctor/M and M pharmaceuticals and Sabinsa pharmaceuticals).
  Arms: Placebo

SUMMARY:
The researchers are doing this study to look at how butyrate levels change in participants' stool after they are on a- plant-based diet for at least 12 weeks. All participants will have monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM). We will compare how the plant-based diet, omega-3 fatty acid and curcumin supplements, and placebo (an inactive substance that looks like the study supplements) affect butyrate levels in participants' stool.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MGUS or SMM
* If non light chain MGUS/SMM then M spike must be either ≥ 0.2 g/dL or BM PC ≥10% (both not required)
* If light chain MGUS/SMM then involved must be ≥10 mg/dL or BM PC ≥10% (both not required)
* If IgA MGUS/SMM then an IgA level >350 mg/dL and an abnormal immunofixation is required (M spike criteria not required).
* If IgD MGUS/SMM then an IgD level >50 mg/dL and an abnormal immunofixation is required (M spike criteria not required).
* Age ≥18 years
* Willingness to comply with all study-related procedures
* ECOG performance status of 0-3
* Interested in learning to cook plant based recipes

Exclusion Criteria:

* Patients that already follow a whole foods plant based diet (ovo-lacto-vegetarian or processed junk food vegan diets are not excluded)
* Legume allergy
* Severe allergies such as anaphylactic shock to nuts (specifically cashews). Peanuts are not included in the meals.
* Concurrent participation in weight loss/dietary/exercise programs
* Mental impairment leading to inability to cooperate
* Enrollment onto any other therapeutic investigational study concurrently and up to 180 days prior to study start date
* Concurrent pregnancy
* Positive HBV, HCV or HIV PCR test will need to be treated first and once undetectable viral load patients may enroll
* ≥ Grade 2 electrolyte abnormalities as defined by CTCAEv5.0 (need to be resolved before enrolling on study)
* If in the opinion of the investigator there maybe any concerns regarding the ability of the patient to complete the study safely or any contraindications
* Heavy drinker (defined as >2 drinks per day or >14 drinks per week)
* Current self-reported illicit drug use (eg heroin, cocaine not marijuana)
* Plan for prolonged travel during the study that would preclude adherence to prescribed diets
* History of major gastrointestinal surgery (not including appendectomy or cholecystectomy) within 3 months of enrollment
* If already taking curcumin or omega 3 supplements patients must be willing to stop it on the date of trial consent for study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Stool microbiome diversity at 12 weeks | 12 weeks
  To evaluate the change in stool microbiome diversity on a dietary vs supplement vs placebo intervention at 12 weeks when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Urvi A Shah, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Emory University (Data Collection Only), Atlanta, Georgia
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm